CLINICAL TRIAL: NCT03298035
Title: A Comparison of Non-invasive Ventilation Methods Used to Prevent Endotracheal Intubation Due to Apnea in Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Catherine Claire Beaullieu, Neonatal-Perinatal Medicine Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-17-0458
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Results first posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Apnea of Prematurity
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NCPAP as mode for apnea prevention (Active Comparator): With recurrence of apneic events, infants on NCPAP will have changes made in NCPAP settings per the clinical team's discretion in attempt to prevent future apneic events. If apneic events persist despite NCPAP adjustments, clinicians may intubate based on clinical judgment.
  Interventions: Device: NCPAP as mode for apnea prevention
- NIPPV as rescue mode for apnea prevention (Experimental): With recurrence of apneic events, infants will be placed on NIPPV with settings and adjustments per the clinical team's discretion. If apneic events persist despite NIPPV placement and setting adjustments, clinicians may intubate based on clinical judgment.
  Interventions: Device: NIPPV as rescue mode for apnea prevention

INTERVENTIONS:
Device: NCPAP as mode for apnea prevention — With recurrence of apneic events, infants on NCPAP will have changes made in NCPAP settings per the clinical team's discretion in attempt to prevent future apneic events. If apneic events persist despite NCPAP adjustments, clinicians may intubate based on clinical judgment.
  Arms: NCPAP as mode for apnea prevention
Device: NIPPV as rescue mode for apnea prevention — With recurrence of apneic events, infants will be placed on NIPPV with settings and adjustments per the clinical team's discretion. If apneic events persist despite NIPPV placement and setting adjustments, clinicians may intubate based on clinical judgment.
  Arms: NIPPV as rescue mode for apnea prevention

SUMMARY:
The purpose of this study is to determine whether nasal intermittent positive pressure ventilation (NIPPV) reduces the need for endotracheal intubation in very low birth weight infants with persistent apnea who fail nasal continuous positive airway pressure (NCPAP).

ELIGIBILITY:
Inclusion Criteria:

* Infants born at < 30 weeks gestational age who develop clinically significant apnea while on NCPAP > 6cm H2O or whose team is considering intubation due to apnea. Consider clinically significant apnea as 1 or more events treated with bag-mask ventilation or 3 episodes of apnea requiring stimulation within 1 hour.
* Infants on maximum caffeine therapy (10mg/kg/day)

Exclusion Criteria:

- Major congenital anomalies including congenital heart disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Beaullieu, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NIPPV as Rescue Mode for Apnea Prevention | NCPAP as Mode for Apnea Prevention
Started | 10 | 9
Received Intervention | 9 | 7
Completed | 9 | 7
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NIPPV as Rescue Mode for Apnea Prevention | NCPAP as Mode for Apnea Prevention | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational age
  weeks | 25.8 (0.8) | 25.8 (2.2) | 25.8 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 3 | 7 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 3 | 4 | 7
  Asian | 2 | 0 | 2
  Causcasian | 1 | 1 | 2
  Hispanic | 4 | 4 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 19
Birth Weight [Mean (Standard Deviation); unit: grams] | 773 (160.5) | 858 (293.4) | 835 (313.3)
Weight at Enrollment [Mean (Standard Deviation); unit: grams] | 920 (286.6) | 921 (204.4) | 920.6 (236.7)
Corrected Gestational Age [Mean (Standard Deviation); unit: weeks] | 28.4 (2.5) | 28.4 (1.1) | 28.4 (2.0)
Number of Participants with Antenatal Glucocorticoid Exposure [Count of Participants; unit: Participants] | 5 | 3 | 8
Number of Participants Who Received Surfactant [Count of Participants; unit: Participants] | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Intubated
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | NIPPV as Rescue Mode for Apnea Prevention | NCPAP as Mode for Apnea Prevention
Number analyzed (Participants) | 10 | 9
Participants | 6 | 8

2. Primary Outcome: Duration of Intubation
Time Frame: 28 days after randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NIPPV as Rescue Mode for Apnea Prevention | NCPAP as Mode for Apnea Prevention
Number analyzed (Participants) | 10 | 9
days | 10.6 (10.2) | 17.5 (11.4)

3. Secondary Outcome: Number of Apneic Events
Time Frame: 28 days after randomization
Population: One participant in the NIPPV group died; therefore, this data was not collected for that participant.
Measure: Mean (Standard Deviation); unit: Number of apneic events
Arm/Group | NIPPV as Rescue Mode for Apnea Prevention | NCPAP as Mode for Apnea Prevention
Number analyzed (Participants) | 9 | 9
Number of apneic events | 3.78 (3.42) | 6.22 (5.52)

4. Secondary Outcome: Number of Participants With Bronchopulmonary Dysplasia (BPD)
Time Frame: 36 weeks corrected gestational age
Population: One participant in the NIPPV group died; therefore, this data was not collected for that participant.
Measure: Count of Participants; unit: Participants
Arm/Group | NIPPV as Rescue Mode for Apnea Prevention | NCPAP as Mode for Apnea Prevention
Number analyzed (Participants) | 9 | 9
Participants | 9 | 8

5. Secondary Outcome: Number of Participants With Necrotizing Enterocolitis (NEC)
Time Frame: 36 weeks corrected gestational age
Population: One participant in the NIPPV group died; therefore, this data was not collected for that participant.
Measure: Count of Participants; unit: Participants
Arm/Group | NIPPV as Rescue Mode for Apnea Prevention | NCPAP as Mode for Apnea Prevention
Number analyzed (Participants) | 9 | 9
Participants | 1 | 5

6. Secondary Outcome: Number of Participants With Air Leak Disorders
Description: Air leak disorders include pneumothorax and/or pneumomediastinum.
Time Frame: 36 weeks corrected gestational age
Population: One participant in the NIPPV group died; therefore, this data was not collected for that participant.
Measure: Count of Participants; unit: Participants
Arm/Group | NIPPV as Rescue Mode for Apnea Prevention | NCPAP as Mode for Apnea Prevention
Number analyzed (Participants) | 9 | 9
Participants | 0 | 0

7. Secondary Outcome: Weight Gain
Time Frame: 36 weeks corrected gestational age
Population: Data were not collected for this outcome measure.
Arm/Group | NIPPV as Rescue Mode for Apnea Prevention | NCPAP as Mode for Apnea Prevention
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Length of Hospital Stay
Time Frame: about 10 to 18 weeks
Population: One participant in the NIPPV group died; therefore, this data was not collected for that participant.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NIPPV as Rescue Mode for Apnea Prevention | NCPAP as Mode for Apnea Prevention
Number analyzed (Participants) | 9 | 9
days | 136 (57.7) | 149 (67.1)

9. Secondary Outcome: Number of Participants Who Died
Time Frame: until discharge (about 10 to 18 weeks) or death
Measure: Count of Participants; unit: Participants
Arm/Group | NIPPV as Rescue Mode for Apnea Prevention | NCPAP as Mode for Apnea Prevention
Number analyzed (Participants) | 10 | 9
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 28 days. Serious and other adverse events were considered as those specifically occurring during the 28-day intervention period; however, mortality was evaluated over the maximum of an 18 week duration. The patient death that occurred happened to be within the 28-day study period.
Arm/Group | NIPPV as Rescue Mode for Apnea Prevention | NCPAP as Mode for Apnea Prevention
All-Cause Mortality (participants affected / at risk) | 1/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

LIMITATIONS AND CAVEATS:
This was a pragmatic trial with inherent bias, as blinding was not possible. There was a small sample size (intent was to enroll 50, but only a few of all screened qualified for escalation of care).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT03298035/Prot_SAP_000.pdf